CLINICAL TRIAL: NCT04297566
Title: MICISPORT Patient Questionnaire
Brief Title: MICISPORT Survey : Questionnaire
Acronym: MICISPORT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL20_0027
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2020-07-29 (Actual); Status verified 2020-07

CONDITIONS: Crohn's Disease
Keywords: disease activity; eating habits; sport; physical activity
MeSH Terms: conditions — Crohn Disease; Feeding Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Crohn disease's patients: Crohn's disease patients seen in gastroenterology consultation or coming in day hospital for treatment

SUMMARY:
This study offers a questionnaire to patients with Crohn's disease in order to assess their physical activity and / or sport as well as their eating habits in order to assess the impact of these lifestyle habits on activity and the symptoms of the disease.

DETAILED DESCRIPTION:
This questionnaire, validated with Doctor Pineton de Chambrun, is set up within the framework of an exercise thesis in pharmacy focusing on the impact of physical activity and diet on the evolution and patients' Crohn's disease (CD) experience. Along with ulcerative colitis (UC), Crohn's disease belongs to chronic inflammatory bowel disease (IBD), which is a major public health concern. These pathologies currently affect 2.5 million patients in Europe (1 million of CD versus 1.5 million of UC). More specifically, in France in 2015, there were 212,700 patients with IBD, with a proportion of 60% CD and 40% RCH1. These pathologies have a major impact on patient's lifes, both in terms of quality of life and the therapeutic course (efficacy and side effects).

Physical activity and diet are other important concerns of health authorities. They are the subject of numerous recommendations based on age and health status. The World Health Organization (WHO), for example, recommends that adults between the ages of 18 and 64 should practice endurance physical activity of moderate intensity lasting at least 150 minutes per week or 75 minutes per day, sustained intensity endurance activity, or a combination of these two types of activity. Epidemiological data show that the lack of physical activity and a sedentary lifestyle favor the increase of the prevalence of diseases, such as cancer and diabetes, but also the increase in cardiovascular risk factors, such as hypertension, obesity and hyperglycemia. A sedentary lifestyle is also considered to be the fourth risk factor for mortality worldwide. Therefore, it appears interesting to study the potential impact of physical activity and exercise as well as food consumption on the activity of Crohn's disease. This impact felt by patients will be assessed by means of a questionnaire which will be offered to them after their medical consultation. The hypothesis of this work is that physical activity and / or sports and diet control improve the quality of life for patients with Crohn's disease.

ELIGIBILITY:
Inclusion criteria:

- Crohn's disease patients

Exclusion criteria:

- Patients without Crohn's disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Any patient with Crohn's disease, seen in consultation
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Disease activity/expression | 1 day
  Disease activity/expression on a scale of 0 to 10 (0 corresponding to no symptoms experienced and 10 corresponding to the zenith of the symptomatology). When analysing the questionnaire

SECONDARY OUTCOMES:
Lived pathology | 1 day
  Lived pathology on a scale of 0 to 10 (0 corresponding to the worst experience and 10 to the best). When analysing the questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume BOUTA, Resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC